CLINICAL TRIAL: NCT01192490
Title: Topical Lidocaine on the Cervix and Intra-Cervical Prior to Insertion of Intrauterine Devices
Acronym: 10-053
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Tennessee (Other)
Responsible Party: Terry Williams, DO, University of Tennessee Chattanooga Department of Obstetrics and Gynecology
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 00002301
Record Dates: First submitted 2010-08-26; First posted 2010-09-01 (Estimated); Last update posted 2011-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Contraception
MeSH Terms: interventions — Lidocaine; Levonorgestrel; Lubricants

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lidocaine Arm (Experimental): This arm will receive intracervical and cervical lidocaine prior to placement of a Mirena.
  Interventions: Drug: Lidocaine
- Lubricant (Placebo Comparator): Subjects in this arm will receive KY gel intracervically and on the cervix prior to placement of a Mirena.
  Interventions: Drug: Lubricant

INTERVENTIONS:
Drug: Lidocaine — 5cc of 2% Lidocaine gel will be placed on the cervix and intra-cervically prior to placement of a Mirena
  Other Names: Mirena
  Arms: Lidocaine Arm
Drug: Lubricant — KY Gel will be placed on the cervix and intra-cervically prior to placement of the Mirena
  Other Names: KY gel
  Arms: Lubricant

SUMMARY:
The hypothesis of this study is that topical cervical and intra-cervical lidocaine will decrease pain associated with the insertion of a Mirena® (levonorgestrel intrauterine device).

1. Primary Aim- Determine if topical lidocaine intra-cervically and on the cervix decreases the pain associated with insertion of a Mirena® (levonorgestrel intrauterine device).

DETAILED DESCRIPTION:
There have been multiple studies performed to determine a medication that will decrease the pain associated with intrauterine device insertion. These studies have tested the use of misoprostol as well as NSAIDS to determine if these decrease the pain associated with insertion. There has also been one small, poorly performed, study that tested the use of intracervical topical lidocaine prior to IUD insertion. Misoprostol and NSAIDS were found to be non-efficacious in decreasing pain. Topical lidocaine was shown to be effective, however, secondary to this being a poorly performed study, additional studies are needed. This study is to determine if topical lidocaine does indeed decrease the pain associated with insertion of the Mirena® (levonorgestrel intrauterine device).

This is a double blinded experimental study to determine whether or not topical lidocaine gel applied to the cervix and intra-cervically decreases pain associated with insertion of the Mirena® (levonorgestrel intrauterine device). Subjects will be randomized into two groups. One group will receive 2% lidocaine gel on the cervix and intra-cervically. The other group will receive a placebo, which will consist of KY being placed on the cervix and intra-cervically. After the Mirena® (levonorgestrel intrauterine device) is inserted, each subject's pain will be assessed by using a visual analog pain scale, and their response will be recorded on the information form. This pain scale will be assessed at the time of insertion, five minutes after insertion, and ten minutes after insertion. The only other study that researched the use of topical lidocaine prior to insertion of an IUD only recorded a pain scale at the time of insertion. Additional scores will be recorded at five and ten minutes to determine if pain is reduced in those time periods. These time periods have been chosen in order that all of this information can be recorded during a normal office visit. A visual analog pain scale is the scale included which measures pain on a scale of zero to ten with zero being no pain at all and ten being the worst pain of your life. This pain scale will be a scale ranging from zero to ten with faces depicting the amount of pain involved for each score. Since there will be different physicians placing the intrauterine devices, there will be a protocol on how to perform the insertion in an attempt to make all insertions as uniform as possible. A copy of this protocol has been included.

ELIGIBILITY:
Inclusion Criteria:

1. Any subject receiving a Mirena® (levonorgestrel intrauterine device) for standard indications.
2. Subjects who received nonsteroidal anti-inflammatory drugs (NSAIDS) will not be excluded.

Exclusion Criteria:

1. Subjects do not desire to be involved in the study
2. Subjects who have taken narcotics.
3. If the Mirena® (levonorgestrel intrauterine device) is not able to be successfully placed.
4. If cervical dilation is required, these subjects will be placed in a separate subset and will be reported on separately.
5. Subject has allergy to lidocaine.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2010-08; Primary Completion 2012-09 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Determine if topical lidocaine intra-cervically and on the cervix decreases the pain associated with insertion of a Mirena® (levonorgestrel intrauterine device). | 2-3yrs
  In order to analyze the data, pain scores will be stratified into three different categories. These categories will be as follows: visual analog scale (VAS) score of 0-2, VAS score of 2-4, VAS score of 5 and greater. This will allow an odds ratio to be calculated and the use of a Chi Square analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Kirk Brody, MD, Principal Investigator — University of Tennessee Chattanooga Department of Obstetrics and Gynecology
Locations (1):
- University of Tennessee Chattanooga Department of Obstetrics and Gynecology, Chattanooga, Tennessee, United States